CLINICAL TRIAL: NCT03883958
Title: Comparison of Thoracic Erector Spinae Plane Block With Thoracic Paravertebral Block for Pain Management in Patients With Unilateral Multiple Fractured Ribs
Brief Title: Erector Spinae Plane Block vs Paravertebral Block for Pain Management in Fractured Ribs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelhamid Youssef Ahmed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESPB vs. TPVB in Rib Fractures
Record Dates: First submitted 2019-03-14; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Rib Fracture Multiple

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPVB (Active Comparator)
  Interventions: Procedure: Paravertebral Block
- ESPB (Experimental)
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — ESPB will be performed in sitting or lateral decubitus position. The target vertebral level will be correspond to the approximate mid-point of the extent of fractured ribs. The tip of the transverse process of the target vertebra will be identified using the high-frequency linear placed in cephalocaudal orientation about 3 cm to the spinous process. The skin and subcutaneous tissue will be infiltrated with 2-3 ml of 2% lignocaine. With the transducer fixed over the targeted TP, a 22-gauge 88-mm needle (Spinocan, B. Braun, Germany) will be advanced in-plane to the ultrasound beam in a cephalo-caudal direction to contact the TP. Correct needle tip position will be confirmed by doing alternating aspiration to confirm lack of inadvertent vascular puncture with injection of 1-2 ml of saline and visualizing linear fluid spread deep to erector spinae muscle, separating it from the TP. A bolus dose (2ml/segment) of plain bupivacaine 0.5% plus 4mg of Dexamethasone will be injected.
  Arms: ESPB
Procedure: Paravertebral Block — TPVB will be performed at a spinal level midway between the uppermost and the lowest fractured rib with the patient in sitting or lateral decubitus position (with patients lying on their unaffected side). The ultrasound-guided technique will be used. A high-frequency linear transducer will be used to confirm the levels of the fractured ribs. The most cephalad and most caudad fractured ribs will be identified first. The fractured rib in the middle will be then identified, and the rib will be then traced back medially. After skin and subcutaneous tissue infiltration with 2-3 ml of 2% lignocaine, a 22-gauge 88-mm needle (Spinocan, B. Braun, Germany) will be inserted in a lateral-to-medial direction until the needle tip entered the paravertebral space. 1-2 ml of Saline will be injected into the paravertebral space while observing the pleura being moved deeply. A bolus dose (2ml/segment) of plain bupivacaine 0.5% plus 4mg of Dexamethasone will be injected.
  Arms: TPVB

SUMMARY:
Rib fractures pose a significant healthcare burden with its associated morbidity, long term disability, and mortality. Pulmonary morbidity is increased in these patients as a result of diminished gas exchange from fracture induced pulmonary injury and from inadequate analgesia compromising both ventilation and pulmonary mechanics. Adequate analgesia is paramount in enhancing pulmonary hygiene aimed at preventing atelectasis and pneumonia. Numbing the nerves to the fractured ribs by injecting local anaesthetic (LA) improves breathing and reduces the risk of complications. Two techniques of regional anesthesia (erector spinae plane block (ESPB) and paravertebral block (PVB)) will be compared regarding their efficacy for treating pain caused by rib fractures. The LA is injected near nerves at two different locations. The PVB is immediately adjacent to the vertebrae, whereas the ESPB is slightly further away from the midline. Both techniques use ultrasound to ensure the LA is directed to the intended place. Adult patients with > 3 consecutive fractured ribs will be consented, then randomised to receive either a ESPB or a PVB. It is expected that both groups will significantly improve in terms of pain score, opioids need, and breathing ability, however it is unclear which technique will provide better results and less complications.

DETAILED DESCRIPTION:
Rib fractures occur most commonly because of blunt thoracic trauma and occur in up to 12% of all trauma patients. Rib fractures themselves pose a significant healthcare burden with its associated morbidity, long term disability, and mortality. Pulmonary morbidity is increased in these patients as a result of diminished gas exchange from fracture induced pulmonary injury and from inadequate analgesia compromising both ventilation and pulmonary mechanics. Various factors affect outcome and mortality after rib fractures. These include the number of ribs fractured, preexisting comorbidities, advanced age, and level of associated pain. Of these, pain is a significant modifiable factor.

Adequate analgesia is paramount in enhancing pulmonary hygiene aimed at preventing atelectasis and pneumonia. Systemic analgesia is usually sufficient in younger patients with fewer undisplaced fractures without a flail segment. Regional techniques are particularly useful in elderly patients (>65 years of age), patients with multiple rib fractures (MRFs), and in patients with severe pain or compromised pulmonary function. Conventional regional techniques used to manage rib fractures include epidural analgesia, paravertebral block (PVB), intercostal, and intrapleural block.

In 2010 Truitt et al. introduced a novel technique whereby local anesthetic (LA) infiltration superficial to the posterior ribs via tunneled catheters successfully controlled rib fracture pain. Since then, multiple thoracic RA (Regional Anesthesia) techniques have been developed that use ultrasound-guided (USG) LA (local anesthetic) injections into fascial planes from the thoracic spinal lamina to the sternum to anesthetize various regions of the thorax.

Some of the conventional regional techniques, particularly epidural analgesia and PVB, may not be feasible in the presence of anticoagulation, multisystem trauma, or in patients unable to be optimally positioned. Recently, several ultrasound-guided (USG) myofascial plane blocks (both single injection and continuous catheter techniques) have been described (e.g. The serratus anterior plane (SAP) block and the erector spinae plane (ESP) block) , which offer the advantages of being less invasive technique and provide adequate analgesia after rib fractures.

ESP block is a novel myofascial plane block recently introduced into clinical practice. It has been successfully utilized in the management of pain after both rib fractures and surgery of the abdomen and thorax, and in the management of chronic thoracic pain. In contrast to the SAP block, the ESP block has the ability to provide analgesia to both the anterior and posterior hemithorax, making it particularly useful in the management of pain after extensive thoracic surgery or trauma (anterior, lateral, and posterior chest wall). Innervation of the ribs and adjoining tissue is primarily through thoracic spinal nerves. After emerging from the spinal cord and traversing through the intervertebral foramina, the thoracic spinal nerves split into ventral and dorsal rami. The ventral rami continue as intercostal nerves innervating the lateral and anterior chest wall, whereas the dorsal rami innervate the posterior chest wall after exiting the paravertebral space.

The ESP block is directed at the erector spinae myofascial plane, which is located on the posterior chest wall between the anterior surface of the erector spinae muscle and oriented cephalocaudally to the posterior surface of the spinal transverse process. Local anaesthetic injected in this plane can block the dorsal rami as they traverse the erector spinae plane, producing anesthesia to the posterior hemithorax. Local anaesthetic also spreads anteriorly and cephalocaudally in the erector spinae plane. Ventral rami and intercostal nerves are blocked by anterior spread, providing analgesia to ribs and periosteum as well as large cutaneous areas of the lateral and anterior chest wall (by blockade of lateral and anterior branches of the intercostal nerves). Cephalocaudal spread provides anesthesia to at least three segments above and four segments below the injection site; a single injection can result in extensive thoracic anesthesia.

PVB has been shown to be as effective as epidural analgesia in managing multiple rib fractures (MRFs). A recent randomized trial has shown that PVB is superior to intravenous patient-controlled analgesia (IVPCA) in providing better analgesia and improving pulmonary function with MRFs.

Unilateral sensory, motor, and sympathetic block can be achieved when local anaesthetic is injected into the paravertebral space. As this space communicates with the intercostal space laterally and the epidural space medially, a 5-6 dermatome sensory block is possible with a single injection of 20 ml of local anaesthetic. Compared with epidural analgesia, PVB is relatively easy to perform, produces less sympathetic blockade, does not cause urinary retention or pruitis, and allows for an unimpeded neurological assessment. However, there is a small risk for pneumothorax, vascular puncture, pleural puncture and a possibility of toxicity due to the rapid absorption of Local Anaesthetic. TPB can be given by using surface landmarks, nerve stimulator guidance or Ultrasound Guidance (USG). A review suggested that USG blocks are more successful and safe than other techniques.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years old or more.
* Rib Fracture Score 7 or more.
* American Society of Anesthesiologist's physiologic state II-III patients.
* 3-6 consecutive fractured ribs.

Exclusion Criteria:

* Patients who are unable to communicate effectively.
* Sternal fractures.
* Bilateral rib fractures.
* VAS score < 7.
* Preexisting spinal deformity.
* Local sepsis at site of injection.
* Coagulopathy.
* Known allergy to the local anesthetic used in the study.
* Patients having significant trauma outside the chest wall e.g., acute spine or pelvic fracture, severe traumatic brain or spinal cord injury, or abdominal visceral injuries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change in visual pain score | Immediatly before and after intervention, 30 minutes after intervention, 3 hours after intervention, 6 hours after intervention and 24 hours after intervention
  0 meaning no pain at all, and 10 described as the worst pain experienced.
Change in Diaphragmatic excursion | Immediatly before and after intervention, 30 minutes after intervention, 3 hours after intervention, 6 hours after intervention and 24 hours after intervention.
  Normal diaphragmatic excursion should be 3-5 cm, but can be increased in well-conditioned persons to 7-8 cm. This measures the contraction of the diaphragm.
  It is performed by asking the patient to exhale and hold it. The provider then percusses down their back in the intercostal margins (bone will be dull), starting below the scapula, until sounds change from resonant to dull (lungs are resonant, solid organs should be dull). That is where the provider marks the spot. Then the patient takes a deep breath in and holds it as the provider percusses down again, marking the spot where the sound changes from resonant to dull again. Then the provider will measure the distance between the two spots.

SECONDARY OUTCOMES:
Opioid dose used for 24-hour period after the procedure. | 24 hour after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ahmed, Principal Investigator